CLINICAL TRIAL: NCT01979406
Title: A Phase 1 Randomized Double-Blind Positive-Controlled Ascending Dose Study to Evaluate the Safety and Immunogenicity of a Replication-Competent Adenovirus Serotype 4 Anthrax Vector Candidate Vaccines - Ad4-PA (Protective Antigen)and Ad4-PA-GPI (Glycosylphosphatidylinositol)
Brief Title: A Phase 1 Ascending Dose Study to Assess the Safety and Immunogenicity of Adenovirus Anthrax Vector Candidate Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PXVX-PA-100-001
Record Dates: First submitted 2013-10-16; First posted 2013-11-08 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Anthrax Infection
Keywords: Anthrax vaccine
MeSH Terms: conditions — Anthrax | interventions — Anthrax Vaccines; Biothrax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- AVA (Active Comparator): Anthrax Vaccine Adsorbed (0.5 mL) as the placebo control on Days 1, 15 and 29
  Interventions: Biological: AVA
- Ad4-PA-1 (Experimental): Given at 10^9, 10^10 and 10^11 vp
  Ad4-PA at Day 1 + oral placebo on Day 15 + AVA boost at Day 29
  Interventions: Biological: AVA; Biological: Ad4-PA-1
- Ad4-PA-2 (Experimental): Given at 10^9, 10^10 and 10^11 vp
  Ad4-PA at Days 1, 15 and 29
  Interventions: Biological: Ad4-PA-1
- Ad4-PA-3 (Experimental): Ad4 given at 10^9, 10^10 and 10^11 vp
  Ad4 PA-GPI at Day 1 + AVA boost at Day 15 + placebo on Day 29
  Interventions: Biological: AVA; Biological: Ad4-PA-1
- Ad4-PA-GPI-1 (Experimental): Given at 10^9, 10^10 and 10^11 viral particles
  Ad4 PA-GPI at Day 1 + oral placebo on Day 29 + AVA boost at Day 15
  Interventions: Biological: AVA; Biological: Ad4-PA-GPI-1
- Ad4 PA-GPI-2 (Experimental): Given at 10^9, 10^10 and 10^11 viral particles
  Ad4 PA-GPI at Day 1 + placebo on Day 15 + AVA boost at Day 29
  Interventions: Biological: AVA; Biological: Ad4-PA-GPI-1
- Ad4-PA-GPI -3 (Experimental): Given at 10^9, 10^10 and 10^11 viral particles
  Ad4-PA-GPI at Days 1, 15 and 29
  Interventions: Biological: Ad4-PA-GPI-1

INTERVENTIONS:
Biological: AVA — Anthrax Vaccine Adsorbed (0.5 mL) as the placebo control on Days 1, 15 and 29
  Other Names: Anthrax vaccine adsorbed (BioThrax)
  Arms: AVA; Ad4 PA-GPI-2; Ad4-PA-1; Ad4-PA-3; Ad4-PA-GPI-1
Biological: Ad4-PA-1 — Ad4-PA will be given at 10^9, 10^10 and 10^11 on Day, followed by an oral placebo on Day 15 and an AVA boost on Day 29
  Other Names: Adenovirus serotype 4 vector vaccine against anthrax PA
  Arms: Ad4-PA-1; Ad4-PA-2; Ad4-PA-3
Biological: Ad4-PA-GPI-1 — Given at 10^9, 10^10 and 10^11 viral particles
  Ad4 PA-GPI at Day 1 + oral placebo on Day 29 + AVA boost at Day 15
  Other Names: Adenovirus anthrax vaccine serotype 4 against anthrax PA
  Arms: Ad4 PA-GPI-2; Ad4-PA-GPI -3; Ad4-PA-GPI-1

SUMMARY:
The purpose of this study is to evaluate 2 vaccine candidates against anthrax compared to the positive (vaccine) control as studied in normal healthy volunteers.

DETAILED DESCRIPTION:
A Phase 1, randomized, double-blind, positive controlled, increasing dose clinical trial in healthy adult subjects at multiple sites. The study will assess safety and immunogenicity of two adenovirus vaccine candidates against anthrax compared to the positive control, Anthrax Vaccine Adsorbed (AVA). The trial will enroll 108 subjects in the anthrax vector vaccine arms and 12 subjects in the AVA positive control subjects. The study will look at three different dose of oral dosages of Ad4-PA (protective antigen) and Ad4-PA-GPI (10^9, 10^10, 10^11 vp/dose)as well as 3 vaccine administration schedules (1 and 15 days; 1 and 29 days; 1, 15, and 29 days); 2 of 3 schedules will include an intramuscular (IM) AVA booster immunization, 1 schedule will include 3 vaccine administrations of Ad4-PA or Ad4-PA-GPI (glycosylphosphatidylinositol) alone, and 1 schedule will include 3 vaccine administrations of AVA alone.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and give written informed consent.
* Healthy men or women aged 18-40 years old,
* BMI between 18 to 36 kg/m2
* Women of child bearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to vaccination on all vaccination days; they must also be willing to use adequate birth control for the duration of the study and have additional pregnancy tests if indicated.
* Intact upper arms with sufficient muscular tissue in the deltoid region for IM vaccine administration.
* Subject must be available for the study duration
* Subject must avoid strenuous exercise for at least 72 hours prior to each study vaccine administration.

Exclusion Criteria:

* Subject is a healthcare worker who has direct contact with patients or has an household contact (HHC) who is immunodeficient or HIV-positive, pregnant, has an unstable medical condition, or is under the age of 18.
* Subject is a childcare worker or a parent who has direct contact with children 5 years old and younger.
* Subject directly prepares food in the food industry.
* Pregnant or breastfeeding throughout the duration of the study until the final visit
* Military service between 1971 and 1999, or after 2012 when Ad4 vaccine was/is routinely given
* Employment in an industry involved in contact with ruminant animals, veterinary sciences, or other potential exposure to B. anthracis
* Received previous Ad4 vaccination or experimental Ad4 vector vaccines
* Received previous anthrax vaccine
* Received or plans to receive any other approved or investigational vaccines from 30 days prior to the first study vaccination until 30 days after the final study vaccination for live attenuated vaccines and from 15 days prior to the first study vaccination until 15 days after the final study vaccination for inactivated vaccines
* HIV or Hepatitis B or C positive
* Immunodeficient or has an unstable medical condition including psychiatric conditions
* Active or past history of acute or chronic gastrointestinal conditions
* Active or past history of cancer except basal cell carcinoma
* Recipient of bone marrow or solid organ transplant
* Received or plans to receive systemic antiviral medication, within 30 days prior to the first study vaccination
* Known allergy to any component of the study vaccine
* Known allergy to, or known medical condition that precludes use of any systemic antiviral medication
* Received or plans to receive medications indicated for decreasing acidity of stomach including:
* Proton pump inhibitors or antacids or histamine 2-receptor antagonists
* Received or plans to receive immunoglobulin or other blood products within 60 days prior to the first study vaccination
* Received or plans to receive other investigational drugs within 30 days prior to the first study vaccination
* Received or plans to receive systemic immunosuppressive therapy, radiation therapy, or inhaled steroids within 30 days prior to the first study vaccination
* Asthmatic or requires asthmatic medications on a daily basis
* Use of systemic chemotherapy within 5 years prior to study
* Body temperature >38.1°C or acute illness within 3 days prior to vaccination
* History of excessive alcohol consumption, drug abuse, or significant psychiatric illness
* History of Guillain-Barré Syndrome
* Blood donation within 2 months prior to first study vaccination
* Expected to be noncompliant with study visits or plans to move away or be living with different HHCs during the next 8 months
* Drinks more than 1200 mL of tea/coffee/cocoa/cola or other caffeinated beverage per day.
* Any condition or finding that in the view of the primary investigator would impede full study participation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The safety, tolerability and immunogenicity of the Ad4 PA and Ad4 PA GPI vaccines across a range of dosages and schedules. | Day 1 through Day 211
  Safety will be measured by looking at safety labs, Adverse Events (AEs) and vaccine reactogenicity data from Baseline through Day 211. Immunogenicity will be measured by the peak serum antibody response to the PA transgene defined as the highest toxin-neutralizing antibody (TNA) titer achieved by a subject at any time between the first post-vaccination visit though Day 85 (and Day 211 if Day 85 is positive).

SECONDARY OUTCOMES:
Antibody response of the Ad4-PA formulation to Ad4 PA GPI | Day 1 through Day 85 (Day 211 if Day 85 is positive)
  Antibody response will be tested via enzyme-linked immunosorbent assay (ELISA) and the peak PA-ELISA titer defined as the highest ELISA titer achieved by a subject at any time between the first post-vaccination visit and Day 85
Antibody response of the Ad4-PA and Ad4-PA-GPI vaccination regimens to the anticipated AVA PEP regimen. | Days 1 through 85 (Day 211 if Day 85 is positive)
  Antibody response will be tested via ELISA and the peak PA-ELISA titer defined as the highest ELISA titer achieved by a subject at any time between the first post-vaccination visit and Day 85.
Antibody response induced by 3 different dosages of Ad4 PA and Ad4 PA GPI. | Days 1 through 85 (Day 211 if Day 85 is positive)
  Antibody response will be tested via ELISA and the peak PA-ELISA titer defined as the highest ELISA titer achieved by a subject at any time between the first post-vaccination visit and Day 85 and titers will be compared across the 3 different dosages of Ad4 PA and Ad4 PA GPI (10^9, 10^10, 10^11).
TNA and antibody response induced by Ad4 PA and Ad4 PA GPI on 3 different vaccination schedules. | Days 1 through 85 (Day 211 if Day 85 is positive)
  Antibody response will be tested via ELISA and the peak PA-ELISA titer defined as the highest ELISA titer achieved by a subject at any time between the first post-vaccination visit and Day 85, and compared among 3 vaccine schedules:
  1. Day 1: Ad4-PA or Ad4-PA-GPI, Day 15 placebo Day 29 AVA boost;
  2. Day 1:Ad4-PA or Ad4-PA-GPI, Day 15 AVA boost + Placebo; and
  3. Days 1, 15 and 29: Ad4-PA or Ad4-PA-GPI
Pre-existing Ad4 immunity on TNA and PA-ELISA response induced by Ad4 PA and Ad4 PA GPI. | Days 1 through 85 (Day 211 if Day 85 is positive)
  Antibody response will be tested via ELISA and the impact of pre-existing Ad4 serostatus (positive/negative) on TNA and PA-ELISA will be evaluated
Evaluate the kinetics of the TNA and PA-ELISA antibody response induced by 3 different doses of Ad4 PA and Ad4 PA GPI on 3 different administration schedules. | Days 1 through 85 (Day 211 if Day 85 is positive)
  TNA and PA-ELISA titer at each post-vaccination visit as measured by ELISA will be compared across each dose group (10^9, 10^10 and 10^11 vp) and dosing schedule. In addition, the time to peak pre-boost TNA titer and to peak pre-boost PA-ELISA titer will be compared across each dose group and dosing schedule. Cumulative TNA and PA-ELISA seroconversion through each post-vaccination visit and through Day 85
In vivo replication/excretion of the Ad4 PA and Ad4 PA GPI vaccines | Days 1 through 211
  The duration of in vivo replication/excretion will be measured by the Ad4 MN seroconversion and titer measured via ELISA testing. Vaccine take defined as either Ad4 micro-neutralizing (MN) seroconversion and/or detection of vaccine shedding measured by polymerase chain reaction (PCR) and confirmed by culture at any time point from Day 1 through Day 211

OTHER OUTCOMES:
Systemic PA-specific cellular immune response induced by Ad4-PA and Ad4-PA-GPI | Days 1 through 43
  The systemic PA-specific cellular immune response induced by Ad4-PA and Ad4-PA-GPI will be measured via cell-based assay on peripheral blood mononuclear cells(PBMCs). The tests will be performed on Days 1, 15, 29 and 43.
Mucosal PA-ELISA antibody responses induced by Ad4-PA and Ad4 PA-GPI | Days 1 through 29
  PA antibody titers from mucosal samples will be obtained on Days 1 and 29 and titers will be compared among the 2 vaccine candidates.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gurwith, MD, Principal Investigator — Emergent BioSolutions; Jakub Simon, MD, Study Director — Emergent BioSolutions; Mo Elsafy, MD, MSc, Principal Investigator — National Institutes of Health (NIH)
Locations (4):
- United States (4):
  - The Center for Pharmaceutical Research, Kansas City, Kansas
  - Walter Reed Army Institute for Research, Silver Spring, Maryland
  - St. Louis University, St Louis, Missouri
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina